CLINICAL TRIAL: NCT05221983
Title: Vitamin D Level: Reflections of a Public Health Issue in the COVID-19 Pandemic. Does it Affect Mortality and Length of Hospital Stay?
Brief Title: COVID-19 and Vitamin D: Length of Hospital Stay and Mortality
Status: Completed | Type: Observational
Sponsor: Yuksek Ihtisas University (Other)
Collaborators: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Sevan ÇETİN ÖZBEK, Assistant Professor, Yuksek Ihtisas University
Other Study IDs: YuksekIU-SCOZBEK001
Record Dates: First submitted 2022-02-02; First posted 2022-02-03 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: COVID-19 Pandemic; Vitamin D Deficiency
Keywords: COVID-19; Vitamin D; Length of stay; Mortality
MeSH Terms: conditions — COVID-19; Vitamin D Deficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with COVID-19 + with vitamin D levels: Patients with COVID-19 + and vitamin D levels were included in the study retrospectively. Vitamin D level was categorized into 3 groups as inadequacy, deficiency and normal from medical records. No intervention was made.

SUMMARY:
The lack of a pharmacological treatment in the COVID-19 pandemic has pushed scientists to search for this issue. Maintaining optimal health is parallel to adequate and balanced nutrition. In this context, can the protective properties of vitamin D play an important role in this pandemic? brought with it the thought. In this study, it was aimed to examine the effect of vitamin D on mortality and hospital stay in COVID-19 disease.

DETAILED DESCRIPTION:
This research was conducted to examine the effect of vitamin D on mortality and hospital stay in COVID-19 disease. For this, the approval of the Ministry of Health and then the ethics committee was obtained. For this reason, patients with positive PCR tests and hospitalized patients with vitamin D levels in their biochemistry were included in the study.

The data of the patients were obtained from the medical records. Information such as age, gender, comorbidities, length of hospital stay, vitamin D level were included in the study. According to the statistical analyzes obtained from these data, it has been shown that vitamin D level has no effect on mortality and hospital stay in COVID-19 disease.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 PCR (Polymerase Chain Reaction) test positive
* Vitamin D level in biochemical parameters
* Adult patients hospitalized for COVID-19

Exclusion Criteria:

-Patients using drugs that may affect vitamin D absorption, such as corticosteroids, cholesterol-lowering agents, phenobarbital and phenytoin-containing agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with positive COVID-19 PCR (Polymerase Chain Reaction) test and vitamin D level in biochemical parameters, who applied to Ankara City Hospital Neurology-Orthopedics Hospital between 01 August and 31 October 2020.
Sampling Method: Probability Sample
Enrollment: 168 (Actual)
Dates: Start 2021-08-21 (Actual); Primary Completion 2021-11-09 (Actual); Study Completion 2021-11-16 (Actual)

PRIMARY OUTCOMES:
Level of Vitamin D | 1 month later
  Vitamin D levels of patients with a diagnosis of COVID-10. These results were categorized at the level of deficiency/insufficiency/normal.
Relationship between vitamin D level and mortality | 1 month later
  Relationship between survival and death by categorized vitamin D level.
Relationship between vitamin D level and hospital stay | 1 month later
  Length of hospital stay by categorized vitamin D level.

SECONDARY OUTCOMES:
Effects of additional diseases (Diabetes mellitus, hypertension, etc.) on hospital stay and mortality | 1 month later.
  Evaluation of the impact of comorbidities on survival during COVID-19 disease.

CONTACTS AND LOCATIONS:
Overall Officials: Levent Öztürk, MD, Study Director — Republic of Turkey Ministry of Health Ankara City Hospitals Neurology-Orthopedics Hospital
Locations (1):
- Republic of Turkey Ministry of Health Ankara City Hospitals Neurology-Orthopedics Hospital, Ankara, Turkey (Türkiye)